CLINICAL TRIAL: NCT00893581
Title: Multimodal Neuroimaging of Treatment Effects in Adolescent Mania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Melissa Delbello, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: DelBello MM NeuroImaging Study
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Mania; Bipolar Disorder
Keywords: mania; adolescent; bipolar
MeSH Terms: conditions — Mania; Bipolar Disorder | interventions — Quetiapine Fumarate; Lithium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1--Quetiapine & Placebo (Active Comparator): Quetiapine & Placebo in the place of Lithium
  Interventions: Drug: Quetiapine & Placebo
- 2-- Lithium & Placebo (Active Comparator): Lithium & Placebo in the place of Quetiapine
  Interventions: Drug: Lithium and Placebo
- Placebo (Placebo Comparator): Sugar Pill (Placebo) given to mimic drug
  Interventions: Other: Healthy Controls

INTERVENTIONS:
Drug: Quetiapine & Placebo — Bipolar adolescents will be initiated on 100 mg per day of quetiapine (or placebo) and 30 mg/kg (maximum starting dose of 600 mg twice daily) of lithium carbonate (or placebo), depending on randomization assignment. Patients will be given placebo for the medication to which they were not assigned. Quetiapine will be adjusted based on tolerability and response to a target dose of 400-600 mg and lithium will be adjusted to a target dose based on achieving a serum level of 1.0-1.2 mEq/L.
  Arms: 1--Quetiapine & Placebo
Drug: Lithium and Placebo — Bipolar adolescents will be initiated on 100 mg per day of quetiapine (or placebo) and 30 mg/kg (maximum starting dose of 600 mg twice daily) of lithium carbonate (or placebo), depending on randomization assignment. Patients will be given placebo for the medication to which they were not assigned. Quetiapine will be adjusted based on tolerability and response to a target dose of 400-600 mg and lithium will be adjusted to a target dose based on achieving a serum level of 1.0-1.2 mEq/L.
  Arms: 2-- Lithium & Placebo
Other: Healthy Controls — Healthy control (patients given placebo -- sugar pill intended to mimic drug)
  Arms: Placebo

SUMMARY:
Specific Aim 1: To determine the effects of treatment with quetiapine or lithium on brain activation in adolescents. The investigators will use functional magnetic resonance imaging (fMRI) to examine brain activation during an attentional task.

Specific Aim 2: To determine the effects of treatment with quetiapine or lithium on neurometabolite measures, early in their illness course. The investigators will use 1H-MRS to identify myo-inositol (mI), N-acetyl aspartate (NAA), and glutamate (Glu) levels in prefrontal ALN regions.

Specific Aim 3: To determine the relationships among the changes in brain activation and neurometabolite measures, as well as symptomatic improvement in manic adolescents.

DETAILED DESCRIPTION:
Hypotheses 1 & 2 predict that following 6 weeks of treatment with lithium or quetiapine, manic adolescents who demonstrate symptomatic improvement will exhibit normalized (decreased) VLPFC and ACC activation and increased activation of compensatory posterior attentional brain areas as well as normalization of VLPFC and ACC neurometabolite measures (increased NAA and decreased Glu levels) compared with those who do not experience symptomatic improvement and healthy adolescents.

Hypothesis 3 predicts significant associations between fMRI activation changes (i.e. decreased activation in VLPFC and ACC ROIs and increased activation in the posterior attention ROI) and MRS changes (increases in NAA and decreases in Glu levels in the VLPFC and ACC) for patients who exhibit symptomatic improvement with either treatment.

Hypothesis 4 predicts that decreases in mI levels at 1 week will be associated with lithium, but not quetiapine, response at endpoint.

In contrast, Hypothesis 5 predicts higher baseline Cho levels will be associated with quetiapine, but not lithium, response at endpoint.

ELIGIBILITY:
Inclusion/Exclusion Criteria

Inclusion - Bipolar Disorder Subjects:

* DSM-IV-TR12 criteria for bipolar disorder, type I, manic or mixed episode, diagnosed by the Washington University in St. Louis Kiddie Schedule for Affective Disorders and Schizophrenia (WASH-U-KSADS)166,101,102-103,104-105,108
* Baseline YMRS112-114 score > 20;
* Ages 12-17 years 11 months old;
* Fluent in English;
* Provision of written informed consent by a legal guardian and written assent by the subject;
* Tanner scale stages III-V167, in order to include only post-pubescent subjects and minimize brain changes associated with the onset of puberty;168-169
* Less than 2 years from onset of bipolar disorder, defined by age at onset of first DSM-IV-TR affective episode (mania, hypomania, depression or mixed), to establish that our sample is early in their illness course;
* No prior psychiatric hospitalizations, <3 months of lifetime psychotropic medication exposure (with the exception of psychostimulants, since excluding patients with psychostimulant exposure would significantly limit the generalizability of our findings), and no active psychotropic medication during the week (72 hours for psychostimulants and benzodiazepines) prior to the index assessment (no treatment with fluoxetine during the prior month). Please note that patients will NOT be taken off medications for the purpose of this study; instead, this criterion is to exclude subjects receiving treatment at the time of index assessment;
* Does not have a history of intolerance or non-response to lithium or quetiapine;
* Manic or depressive symptoms do not result entirely from acute medical illness or acute intoxication or withdrawal from drugs or alcohol as determined by medical evaluation and rapid symptom resolution;
* No lifetime DSM-IV-TR diagnosis of post-traumatic stress disorder (PTSD), since PTSD has been associated with abnormalities in prefrontal NAA and function170-171,172. Furthermore, bipolar patients with co-occurring PTSD are less likely to respond to lithium monotherapy, and often need a serotonin specific reuptake inhibitor (SSRI) as adjunctive treatment to a mood stabilizer.173,174 ;
* If female and of child bearing potential, agrees to use one of the following method of birth control: complete abstinence from sexual intercourse, barrier (diaphragm or condom), or oral/injectable contraceptive.

Inclusion - Healthy Controls:

* Ages of 12-17 years and 11 month;
* No history of any DSM-IV-TR Axis I disorder (nicotine dependence is permitted);
* No first- or second-degree relatives with an affective or psychotic disorder;
* No medications with central nervous system effects within 5 half-lives;
* Fluent in English;
* Tanner stage III-V;
* Provision of informed consent and assent.

Exclusion - Bipolar Subjects & Healthy Controls:

* Contraindication to an MRI scan (e.g., braces or claustrophobia);
* An unstable medical or neurological illness that could influence fMRI or MRS results;
* IQ < 70, as determined by The Wechsler Abbreviated Scale of Intelligence (WASI) ;
* A positive pregnancy test;
* A history of major medical or neurological illness or a significant episode (> 10 minutes) of loss of consciousness;
* Any lifetime DSM-IV-TR substance use disorder (nicotine dependence is permitted);
* A lifetime DSM-IV-TR diagnosis of any pervasive developmental disorder;
* The patient lives >100 miles from the University of Cincinnati or is not able to attend follow-up visits.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2009-03; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to use magnetic resonance imaging (MRI) to examine brain structure, function and chemistry in people with Bipolar I disorder (manic or mixed episodes) who are being treated with either quetiapine or lithium. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Melissa DelBello, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lei D, Li W, Qin K, Ai Y, Tallman MJ, Patino LR, Welge JA, Blom TJ, Klein CC, Fleck DE, Gong Q, Adler CM, Strawn JR, Sweeney JA, DelBello MP. Effects of short-term quetiapine and lithium therapy for acute manic or mixed episodes on the limbic system and emotion regulation circuitry in youth with bipolar disorder. Neuropsychopharmacology. 2023 Mar;48(4):615-622. doi: 10.1038/s41386-022-01463-6. Epub 2022 Oct 13. PMID 36229596
- [Derived] Li W, Lei D, Tallman MJ, Ai Y, Welge JA, Blom TJ, Fleck DE, Klein CC, Patino LR, Strawn JR, Gong Q, Strakowski SM, Sweeney JA, Adler CM, DelBello MP. Pretreatment Alterations and Acute Medication Treatment Effects on Brain Task-Related Functional Connectivity in Youth With Bipolar Disorder: A Neuroimaging Randomized Clinical Trial. J Am Acad Child Adolesc Psychiatry. 2022 Aug;61(8):1023-1033. doi: 10.1016/j.jaac.2021.12.015. Epub 2022 Jan 25. PMID 35091050
- [Derived] Patino LR, Klein CC, Strawn JR, Blom TJ, Tallman MJ, Adler CM, Welge JA, DelBello MP. A Randomized, Double-Blind, Controlled Trial of Lithium Versus Quetiapine for the Treatment of Acute Mania in Youth with Early Course Bipolar Disorder. J Child Adolesc Psychopharmacol. 2021 Sep;31(7):485-493. doi: 10.1089/cap.2021.0039. Epub 2021 Sep 14. PMID 34520250